CLINICAL TRIAL: NCT00671632
Title: A Randomized, Single Center, Double-Blind, Multiple-Dose, Placebo-Controlled, Crossover, Double-Dummy Study of The Acute Behavioral and Subjective Effects of Ramelteon in Subjects With a History of Polydrug Abuse.
Brief Title: Behavioral and Subjective Efficacy of Ramelteon in Subjects With a History of Polydrug Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-015; U1111-1114-3109 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Drug Abuse
Keywords: Addiction
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — ramelteon; Triazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramelteon, triazolam, and placebo (56 poss. combinations) (Experimental): Ramelteon, triazolam, and placebo (56 possible combinations total)
  Interventions: Drug: Ramelteon, triazolam, and placebo (56 possible combinations total)

INTERVENTIONS:
Drug: Ramelteon, triazolam, and placebo (56 possible combinations total) — Randomized sequence over eight consecutive days to include the following:
  Ramelteon 16 mg, tablets, orally, one day only;
  Ramelteon 80 mg, tablets, orally, one day only;
  Ramelteon 160 mg, tablets, orally, one day only;
  Triazolam 0.25 mg, capsules, orally, one day only;
  Triazolam 0.50 mg, capsules, orally, one day only;
  Triazolam 0.75 mg, capsules, orally, one day only;
  Ramelteon placebo-matching tablets, orally, one day only, OR Triazolam placebo-matching capsules, orally, one day only;
  Additional dose of study medication or placebo, tablets or capsules, orally, one day only.
  Other Names: Rozerem™; TAK-375

SUMMARY:
The purpose of this study is to determine the relative abuse potential of ramelteon, once daily (QD), compared to triazolam in subjects with a history of drug abuse.

DETAILED DESCRIPTION:
Insomnia is characterized by a complaint of either difficulties initiating and maintaining sleep, or of nonrestorative and non-refreshing sleep. Transient insomnia affects approximately one-third to one-half of the US population, based on the results of 2 surveys of representative samples of the adult US population conducted by the Gallup Organization in which respondents were asked if they had "ever had difficulty sleeping." Based on reports of "regular" or "frequent" sleep difficulty, results from the same studies suggest that approximately one-tenth of the US population experiences chronic insomnia. The ideal treatment for insomnia would reduce the latency to onset of sleep and increase total sleep time, without a negative impact on sleep architecture and without safety concerns or next-day effects.

Ramelteon is a melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

Participation in this study is anticipated to be about 1 month.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Must be in good health as determined by a physician (ie, via medical history and physical examination).
* Clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory unless the results are deemed not clinically significant by the investigator or sponsor.
* Must have a history of substance abuse or dependence, on a commonly abuse recreational psychoactive drug (e.g., benzodiazepines, cocaine, opiates, cannabinoids).
* Must have a negative urine sample for substances of abuse and a negative breathalyzer test before the first dose of study medication is administered.
* Must be free of any signs/symptoms of withdrawal from substances after admittance to the research unit and prior to the first dose of study medication.
* Must report liking for study medication given on Day -2 and liking must be of greater magnitude that than the liking for study medication given on Day -1.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds including melatonin.
* Known hypersensitivity to benzodiazepines or related compounds.
* Current diagnosis of any type of physical drug dependence other than nicotine or caffeine.
* Positive HBsAg are excluded.
* Positive human immunodeficiency virus antibody at screening.
* Diastolic blood pressure greater than 90 mm Hg or a systolic pressure of greater than 140 mm Hg at screening.
* Previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study drug.
* Body weight is less than 99 or greater than 264 pounds. Subjects that are morbidly obese as defined by greater than 2 times ideal body weight
* Significant urine concentration of any drug that could interfere with the study.
* Clinically significant abnormal finding on physical examination or electrocardiogram. Subjects with a clinically significant illness in the past 30 days.
* Current Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised diagnosis of a serious psychiatric condition (e.g. Schizophrenia, Major Depression).
* Currently is participating in another investigational study or has participated in an investigational study within the past 30 days.
* Any other serious disease or condition at screening or at randomization that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2003-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Peak liking score from the Drug Effect Questionnaire as recorded during the 24 hours following administration. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit

SECONDARY OUTCOMES:
Next Day Questionnaire. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Addiction Research Center Inventory. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Drug Effect Questionnaire. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Subjective Effects Questionnaire. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Pharmacologic Class Questionnaire. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Drug Versus Money Multiple Choice Procedure. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Observer Rated Questionnaire. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Word Recall/Recognition Task. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Enter and Recall Task. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Balance task. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Digit Symbol Substitution Task. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Circular lights task. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Neuropsychometric Testing | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Adverse Events | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Laboratory Test Results | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Vital Signs | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Electrocardiograms | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit
Physical Examination Findings. | Days 1, 2, 3, 4, 5, 6, 7, and 8 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- [Result] Johnson MW, Suess PE, Griffiths RR. Ramelteon: a novel hypnotic lacking abuse liability and sedative adverse effects. Arch Gen Psychiatry. 2006 Oct;63(10):1149-57. doi: 10.1001/archpsyc.63.10.1149. PMID 17015817
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI